CLINICAL TRIAL: NCT06638541
Title: Dose dE-eScalaTion IN prostATe radIOtherapy usiNg an MR-Linac in 2 Fractions - a Randomised Trial
Brief Title: Dose dE-eScalaTion IN prostATe radIOtherapy usiNg an MR-Linac in 2 Fractions
Acronym: DESTINATION 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Elekta Limited (Industry); MRL Consortium (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR5984; 338368 (Other: IRAS)
Record Dates: First submitted 2024-09-23; First posted 2024-10-15 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: De-escalation; Radiotherapy; MR-Linac
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Uniform dose (Active Comparator): Arm 1 (Uniform dose) will receive 27 Gy in 2 fractions to the whole prostate + seminal vesicles (SV), the CTV, with 0 mm CTV-PTV margin.
  Interventions: Radiation: Prostate radical radiotherapy
- De-escalated dose (Experimental): Arm 2 (De-escalated dose) will use two dose levels:
  The benign prostate (on MRI) will receive 20 Gy in 2 fractions with a 0mm PTV margin.
  The intraprostatic tumour mass(es) as seen on MRI will receive 27 Gy in 2 fractions. A 4mm GTV-PTV margin will be added to the MR visible tumour to form PTV 27Gy.
  Interventions: Radiation: Prostate radical radiotherapy

INTERVENTIONS:
Radiation: Prostate radical radiotherapy — Radiation: De-escalated radiotherapy to be delivered on the Elekta Unity MR-linac

SUMMARY:
DESTINATION 2 is a multi-centre randomised trial treating intermediate risk localised prostate cancer with 2 fraction Stereotactic Body Radiotherapy (SBRT). All radiotherapy will be delivered in two fractions (sessions) on an MR Linac using daily adaptation. Men will either receive uniform dose radiotherapy or de-escalated dose radiotherapy. The primary endpoint is acute GU CTCAE v5 grade 2+ toxicity. It will also look at late toxicity, patient-reported outcome measures and PSA control.

DETAILED DESCRIPTION:
54 patients meeting inclusion criteria will be randomised between two arms. Arm 1 (Uniform dose) will receive 27 Gy in 2 fractions to the whole prostate + seminal vesicles (SV), the CTV, with 0 mm CTV-PTV margin. Arm 2 (De-escalated dose) will use two dose levels: The benign prostate (on MRI) will receive 20 Gy in 2 fractions with a 0mm PTV margin. The intraprostatic tumour mass(es) as seen on MRI will receive 27 Gy in 2 fractions. A 4mm GTV-PTV margin will be added to the MR visible tumour to form PTV 27Gy. The primary endpoint is emergent acute GU CTCAE v5 Grade 2+ toxicity, recorded within 3 months of completing radiotherapy. Secondary endpoints are CT CAE v5 acute GI toxicity, late toxicity, patient-reported outcome measures (PROMs) (EPIC-26, IPSS, and IIEF-5) at 4 and 12 weeks, 6 months, 1 and 2 years post treatment, PSA control and kinetics

ELIGIBILITY:
Inclusion Criteria:

1. Men aged ≥18 years
2. Histological confirmation of prostate adenocarcinoma requiring radical radiotherapy
3. Gleason score 3+3, 3+4 or 4+3 (Grade groups (GG) 1, 2 or 3)
4. MRI stage T3a or less (as staged by AJCC TNM 2018). MRI must be performed within a year of randomisation
5. MRI-visible tumour(s) of PIRADS v2 grade 3 or higher and able to be delineated on T2 and diffusion-weighted imaging +/- dynamic contrast-enhanced imaging. Tumour nodule visible on MRI should be considered able to be boosted by treating clinician and <2.5cm in maximal dimension
6. The MRI-defined lesion must be confirmed as malignant on biopsies (Gleason grade must be within the limits expressed in inclusion factor 3)
7. Patients can be concurrently treated with androgen deprivation therapy (ADT) if this would be standard of care. LHRH analogues, LHRH agonists or Bicalutamide are permitted. ADT is not mandatory where this would usually be omitted.
8. PSA <20 ng/ml prior to starting ADT, if used
9. WHO Performance status 0-2
10. Ability of the participant understand and the willingness to sign a written informed consent form.
11. Willing to consent to contraception during and for 1 year after treatment when applicable.
12. Ability/willingness to comply with the patient reported outcome questionnaires schedule throughout the study.

Exclusion Criteria:

1. Contraindications to MRI (e.g. pacemaker, potentially mobile metal implant, claustrophobia)
2. Severe GU symptoms that would preclude extreme hypofractionation per the discretion of the treating physician.
3. IPSS Score > 19
4. High grade disease (GG3) occult to MRI-defined lesion. As a guide, any pathology for which you would consider surveillance (eg GG1, low volume GG2) is allowed outside of the MRI-defined area.
5. Prostate volume >90cc
6. Comorbidities which predispose to significant toxicity (e.g. inflammatory bowel disease) or preclude long term follow up
7. Hip replacement, or other pelvic metalwork which causes significant artefact on diffusion-weighted imaging
8. Previous pelvic radiotherapy
9. Patients needing >6 months of ADT due to disease parameters.
10. Previous invasive malignancy within the last 2 years where this is likely to shorten lifespan the following will remain eligible: basal or squamous carcinomas of the skin, low risk non-muscle invasive bladder cancer (assuming cystoscopic follow up now negative) or small renal masses on surveillance.
11. Participating in another interventional trial for prostate cancer

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Acute GU toxicity | 12 weeks
  To describe the absolute risk and relative risk reduction of acute genitourinary (GU) toxicity (CTCAE v5) when delivering de-escalated two fraction prostate SBRT compared to uniform dose two fraction prostate stereotactic body radiotherapy (SBRT) for intermediate risk prostate cancer.

SECONDARY OUTCOMES:
Acute Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) toxicity | Baseline, last fraction, week 2, 4 and 12
  To describe the absolute and relative risk of toxicity
Late Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0) toxicity | Month 6, 12, 24
  To describe the absolute and relative risk of toxicity
Feasibility of radiation delivery | At time of treatment
  Feasibility- estimate percentage of fractions interrupted due to patient discomfort
Dosimetry | At time of treatment
  Dosimetry- estimate the accumulated dose differences between the de-escalated and uniform dose delivery
Patient reported outcome measures | Baseline, last fraction of treatment, week 2, 4 and 12, 6 months, 1 and 2 years post treatment.
  To assess baseline, acute and late International Prostate Symptom Score (IPSS). IPSS ranges from 0 to 35. Lower scores are better: A lower score indicates fewer or less severe urinary symptoms, while a higher score suggests more severe symptoms.
Patient reported outcome measures | Baseline, 4 and 12 weeks, 6 months, 1 and 2 years post treatment.
  Expanded Prostate Cancer Index Composite Short Form (EPIC-26). EPIC-26 scores are transformed to a 0-100 scale for each domain.The questionnaire usually covers urinary incontinence, urinary irritative/obstructive symptoms, bowel, sexual, and hormonal functions. Higher scores represent better health-related quality of life.
Patient reported outcome measures | Baseline, 6 months, 1 and 2 years post treatment.
  International Index of Erectile Function-5 (IIEF-5). The IIEF-5 score ranges from 5 to 25. Higher scores are better: A higher score indicates better erectile function, while a lower score suggests more severe erectile dysfunction.
PSA kinetics | Baseline (pre ADT), week 12, month 6, and 1 and 2 years post treatment
  To assess biochemical relapse-free survival at 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alison Tree, Study Chair — Royal Marsden Hospital, Institute of Cancer Research
Locations (2):
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - The Royal Marsden NHS Foundation Trust, Sutton

IPD SHARING:
Plan to Share IPD: Yes
It is intended that data will be shared within the MOMENTUM collaboration, between centres delivering treatment in the same way as DESTINATION2. Pseudonymised data will be stored within MOMENTUM for at least 5 years. Storage will be cloud based and as the treating centre we will have free access to the data and control over who else can assess it.
Time Frame: 5 years